CLINICAL TRIAL: NCT01483638
Title: A Phase II Study of Axitinib as Maintenance Treatment for Patients With Metastatic Colorectal Carcinoma
Brief Title: Axitinib as Maintenance Treatment in Patients With Metastatic CRC
Acronym: TTD-11-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely closed due to lack of accrual
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTD-11-01; 2011-002384-16 (EudraCT Number)
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Carcinoma
Keywords: duration of disease response; axitinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): axitinib
  Interventions: Drug: axitinib
- control (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: axitinib — 5 mg BID taken orally with food continuously on Day 1 of the study. One cycle corresponds to 28 days.
  Arms: Experimental
Drug: placebo — will be administered orally with the same schedule of axitinib
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the maintenance therapy with axitinib in patients with metastatic colorectal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histological or cytological confirmed colorectal adenocarcinoma with metastatic disease documented on diagnostic imaging studies, not susceptible of radical surgery of metastases, and a low burden of disease.
2. Patients without progressive disease after six months of the standard first line chemotherapy regimen for CRC (5FU or capecitabine ± oxaliplatin or irinotecan ± bevacizumab or cetuximab).
3. Patient must have at least one measurable lesion as defined by modified RECIST criteria.
4. Male or female, age ≥18 years.
5. ECOG performance status of 0 or 1 and life expectancy of ≥12 weeks.
6. Adequate organ function as defined by the following criteria:

   * absolute neutrophil count (ANC) ≥1500 cells/mm3;
   * platelets ≥100,000 cells/mm3.
   * Hemoglobin ≥9.0 g/dL.
   * AST and ALT ≤2.5 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT ≤5.0 x ULN;
   * Total bilirubin ≤1.5 x ULN;
   * Alkaline phosphatase <300U/l
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥50 mL/min;
   * Urinary protein <2+ by urine dipstick. If dipstick is ≥2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours.
7. At least 4 weeks since the end of prior systemic treatment, radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 or back to baseline except for alopecia or neurotoxicity
8. No evidence of pre existing uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
9. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
10. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
11. Willingness and ability to comply with scheduled visits, treatment plans (including willingness to take either AG-013736 or placebo according to randomization), laboratory tests, and other study procedures.

Exclusion Criteria:

1. Gastrointestinal abnormalities including:

   * inability to take oral medication;
   * requirement for intravenous alimentation;
   * prior surgical procedures affecting absorption including total gastric resection;
   * treatment for active peptic ulcer disease in the past 6 months;
   * active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
   * malabsorption syndromes.
   * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to start, unless affected area has been removed surgically
2. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine).
3. Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
4. History of haemorrhage within the past 6 months, including gross hemoptysis or hematuria.
5. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
6. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
7. A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
8. Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
9. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females.
10. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
11. History of a malignancy (other than colorectal cancer) except those treated with curative intent for skin cancer (other than melanoma), in situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
12. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
13. Female patients who are pregnant or lactating, or men and women of reproductive potential not willing or not able to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for 6 months after discontinuing study treatment. The definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate.
14. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
15. Current, recent (within 4 weeks of the study treatment administration), or planned participation in an experimental therapeutic drug study other than this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 4 years

SECONDARY OUTCOMES:
overall survival | 4 years
overall response rate | 4 years
duration of disease response | 4 years
Adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Grávalos, MD, Study Chair — Hospital 12 de Octubre; Alfredo Carrato, MD, PhD, Study Chair — Hospital Universitario Ramon y Cajal
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy, Madrid, Madrid, Spain

REFERENCES:
- See also: Related info — http://www.ttdgroup.org